CLINICAL TRIAL: NCT05617287
Title: An Exploratory Investigation of Dietary Supplementation and the Effect on Common Symptoms of Perimenopause and Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semaine Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20265
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Menopause; Menopause Related Conditions; Perimenopausal Disorder
Keywords: Menopause; Perimenopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semaine Supplement (Experimental): Participants are provided with a dietary supplement and are instructed to take 1 capsule per day. Participants are to take the supplement at the same time every day. If forgotten, they are to take it with the next meal. Participants will take a well-being assessment after each month (4 surveys total including the baseline.)
  Interventions: Dietary Supplement: Semaine Menopause Supplement

INTERVENTIONS:
Dietary Supplement: Semaine Menopause Supplement — Synergistic Dietary Supplement

SUMMARY:
A combination of synergistic dietary supplements is hypothesized to significantly improve self-reported measures of menopausal symptoms when compared with a baseline without the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ability to take oral medication and be willing to adhere to the dietary supplement regimen (1 capsule per day)
* Moderate self-reported discomfort related to perimenopause or menopause. Participants will complete the menopause well-being survey and must answer an average of "moderate" or higher.

Exclusion Criteria:

* Current use of medication for high blood pressure or for blood thinning
* Currently undergoing chemotherapy or has previously been treated for cancer
* Pregnancy, breastfeeding, or attempting to become pregnant during the study
* Known allergic reactions to components of the dietary supplement (red clover extract, olive extract, bergamot extract )

Ages: 40 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in perceived discomfort associated with the most common symptoms linked with perimenopause and menopause | 12 weeks
  Symptoms will be reported by the participant on a scale of perceived discomfort and will include rankings for mood, anxiety, fatigue, sleep quality, hot flashes, and libido.
  This survey will be based on the widely used and validated Menopause Rating Scale (MRS). The MRS will be modified to increase dynamic range by changing the response gradations from 5 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, Principal Investigator — Citruslabs; Matthew Crane, Principal Investigator — Semaine Health
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided